CLINICAL TRIAL: NCT04295148
Title: SEQUAR - SEmitendinosus vs QUadriceps in Anterior Cruciate Ligament Reconstruction - a Prospective Randomized Study
Brief Title: SEQUAR SEmitendinosus vs QUadriceps in Anterior Cruciate Ligament Reconstruction
Acronym: SEQUAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Stalman, Senior Consultant, Principal Investigator, Ph.D., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNR 2019-03359
Record Dates: First submitted 2020-02-26; First posted 2020-03-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semitendinosus graft (Active Comparator): Participants receive the Semitendinosus Graft technique during ACL reconstruction.
  Interventions: Procedure: ACL Reconstruction with Semitendinosus graft
- Quadriceps tendon-bone graft (Active Comparator): Participants receive the Quadriceps Tendon-Bone Graft technique during ACL reconstruction.
  Interventions: Procedure: ACL Reconstruction with Quadriceps tendon-bone graft

INTERVENTIONS:
Procedure: ACL Reconstruction with Semitendinosus graft — Participants will undergo Anterior Cruciate Ligament Reconstruction with Semitendinosus graft
  Other Names: ACL-R with Semitendinosus graft; Semitendinosus ACL-R
  Arms: Semitendinosus graft
Procedure: ACL Reconstruction with Quadriceps tendon-bone graft — Participants will undergo Anterior Cruciate Ligament Reconstruction with Quadriceps tendon-bone graft
  Other Names: ACL-R with Quadriceps tendon-bone graft; Quad tendon-bone ACL-R
  Arms: Quadriceps tendon-bone graft

SUMMARY:
Randomized control trial comparing two different Anterior Cruciate Ligament (ACL) grafts in Anterior Cruciate Ligament Reconstruction: the semitendinosus hamstrings graft and the quadriceps graft. Capio Artro Clinic (Stockholm) has vast experience in ACL surgery using both semitendinosus and quadriceps grafts.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the quadriceps graft with bone-plug in Anterior Cruciate Ligament Reconstruction (ACL-R) and compare it with the most common choice of graft, semitendinosus hamstrings graft in ACL-R in athletes with Tegner Activity Scale 7 or higher. Both methods are well-known and continually registered in the Swedish ACL Registry.

Both grafts will be compared post operatively as to knee laxity (primary outcome), PROMs, as well as measure graft site morbidity, Return to Sports rate, and the post-operative rehab. At 9 months we will also preform a MRI scan to determine graft maturity. 5-year and 10-year data will also be acquired through the Swedish ACL-registry and Lysholm score and Tegner Activity Level score. At 10-year a plain weight baring X-ray will be preformed to evaluate development of osteoarthritis.

The study design is a prospective randomized study with equal groups:

Semitendinosus graft (=100) and Quadriceps tendon graft (n=100). According to historical material from Capio Artro Clinic (Stockholm) the following power calculation has been made: Significance lever 5 percent (p=0.05) and power is 80%. The difference between the groups is 1 mm knee laxity with KT-1000 which would give an effect size of 0,44 or less compared to an average effect size (0,50). 85 individuals will be needed in each group in the statistical analysis. Although no stratification for sex will be performed, our aim is to have a balanced representation of sex that reflects the typical patient population for this condition at the clinic, with a distribution of 40% females and 60% males across both groups. Inclusion will continue until we have at least 100 individuals in each group. This means that each group can have more than 100 individuals. Randomization process and study design will be done according to the CONSORT guidelines.

Initially, the study was designed to have two primary outcome measures: KT-1000 knee laxity at 6 months and KOOS at 24 months. However, the study is only powered for the first outcome (Knee Laxity measured with KT-1000), therefore KOOS will be followed as a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Pre-injury Tegner Activity Scale≥7
* Intended return to sports to prior sport and Tegner Activity Scale Level
* Time between injury and inclusion not more than 6 months
* MR verified ACL rupture

Exclusion Criteria:

* Previous knee injury with symptoms before ACL injury
* Neurological disease, inflammatory disease, connective tissue disease or balance disorder
* Previous lower limb fracture or surgery
* Laxity in the medial collateral ligament (MCL) and lateral collateral ligament (LCL) > grade 1
* PCL rupture or Multiligament knee injury (MLKI)
* Radiographic sign of osteoarthritis (OA)
* Previous knee surgery or ligament injury in contralateral knee
* Beighton score ≥ 5

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
KT-1000 Knee Laxity at 6 months | Pre-operative appointment and 6 months post-operative appointments
  The KT-1000 measures laxity objective- and parametrically and is a validated tool for establishing joint laxity post operatively in mm.

SECONDARY OUTCOMES:
KOOS | Pre-operative appointment, 12 months, 24 months, 5 years and 10 years post-operative appointments
  Patients will complete the KOOS at specific time points to evaluate subjective knee function throughout treatment
IKDC | Pre-operative appointment, 12 months, 24 months, 5 years and 10 years post-operative appointments
  Patients will complete the IKDC at specific time points to evaluate subjective knee function throughout treatment.
PAS | Pre-operative appointment, 12 months, 24 months, 5 years and 10 years post-operative appointments
  Patients will complete the PAS at specific time points to evaluate subjective knee function throughout treatment
EQ5D | Pre-operative appointment, 12 months, 24 months, 5 years and 10 years post-operative appointments
  Patients will complete the EQ5D at specific time points to evaluate subjective knee function throughout treatment
Tegner Activity Score | Pre-operative appointment, 6 months, 9 months, 12 months, 18 months, 24 months, 5 years and 10 years post-operative appointments
  Patients will complete the Tegner Activity score at specific time points to evaluate level of sports activity postoperatively.
ACL-RSI | 6 months and 12 months, post-operative appointments
  Patients will complete the ACL-RSI surveys at specific time points to evaluate self efficacy and readiness to return to sports throughout treatment
Return to Sports Questionnaire | 6 months, 9 months and 12 months, 18 months, and 24 months post-operative appointments
  Patients will complete the a Return to Sports Questionnaire at specific time points to evaluate return to sports after 6 and 12 months throughout treatment
Werner anterior knee pain score | 6 weeks, 6 months, 9 months, and 12 months
  Patients will complete Werner anterior knee pain scores at specific time points to evaluate graft site pain/morbidity throughout treatment
Kartus anterior knee pain score | 6 weeks, 6 months, 9 months, and 12 months
  Patients will complete Kartus anterior knee pain score at specific time points to evaluate graft site pain/morbidity throughout treatment
Graft site morbidity questionnaire | 6 weeks, 6 months, 12 months, 24 months
  Patients will complete additional survey questions at specific time points to evaluate graft site pain/morbidity throughout treatment
Goniometric measurement: Knee extension and flexion | 2 weeks, 6 weeks, 6 months, 9 months and 12 months
  Patients will undergo goniometric measurement at specific time points to evaluate knee moment throughout treatment.
Measurement of circumference of the knee | 2 weeks, 6 weeks, 6 months, 9 months and 12 months
  Circumference of the knee will be measured at mid-patella and 15 cm above superior border of the patella. They will be compared with the contralateral knee to compare knee swelling.
Biodex Isokinetic Measurement | 6 months, 9 months and 12 months
  Patients will undergo Biodex Isokinetic measurement at specific time points to muscle strength throughout treatment.
Functional knee tests | 6 months, 9 months and 12 months
  Patients will undergo functional knee test (ie one legged jump and crossover jump) at specific time points to evaluate functional knee movement throughout treatment.
Lachmans test | Pre-operative appointment , 6 months, 9 months and 12 months
  Patients will undergo passive accessory stability tests Lachmans test (graded 0,1,2 and 3) at specific time points to evaluate passive knee laxity throughout treatment.
Pivot shift test | Pre-operative appointment , 6 months, 9 months and 12 months
  Patients will undergo passive accessory stability tests pivot shift test (graded 0,1,2 and 3) at specific time points to evaluate passive knee laxity throughout treatment.
Time to Return to Sports Rates | 6 months, 9 months, 12 months, 18 months, 24 months
  Time to return to sports will be evaluated through Return to Sport surveys at specific time points throughout treatment
Graft failure rate or ACL re-rupture | 10 years
  ACL reconstruction will be evaluated by graft failure rate or ACL re-rupture during a 10 year period
ACL re-operation | 10 years
  ACL reconstruction will be evaluated by re-operation rate during a 10 year period
Graft maturity | 9 months
  Graft maturity after ACL reconstruction will be evaluated by MRI at 9 months postoperatively.
10 year X-Ray | 10 years
  Development of osteoarthritis after ACL reconstruction will be evaluated by plain weight baring X-rays at 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Stålman, MD,PhD, Principal Investigator — Karolinska Institutet; Mikael Östin, MD, Principal Investigator — Capio Artro Clinic AB; Vasileios Sarakatsianos, MD, Principal Investigator — Karolinska Institutet; Joanna Kvist, PhD, Principal Investigator — Karolinska Institutet; Daniel Castellanos, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Capio Artro Clinic AB, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castellanos Dolk D, Sarakatsianos V, Worner T, Ostin M, Cristiani R, Kvist J, Stalman A. Semitendinosus vs quadriceps tendon autograft in anterior cruciate ligament reconstruction (SEQUAR): protocol for a prospective randomized controlled trial. BMC Musculoskelet Disord. 2025 Oct 13;26(1):951. doi: 10.1186/s12891-025-09183-w. PMID 41083992